CLINICAL TRIAL: NCT04077892
Title: A Randomized Trial of Comparing a Combination of Montelukast and Budesonide With Budesonide in Allergic Rhinitis
Brief Title: Compare the Effect of INS Alone and Added LTRA in Treatment of SAR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Luo Zhang, President,Beijing TongRen Hospital, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR-INS&LTRA-AR
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Allergic Rhinitis
Keywords: budesonide; montelukast; combination therapy; monotherapy
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Budesonide; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination of budesonide and montelukast (Experimental): receive treatment with either a combination of budesonide (Rhinorcort Astra Zeneca AB), 1 spray per nostril twice daily (total 256 μg/d) and 10mg oral montelukast tablet (Merck Sharp & Dohme Australia Pty Ltd) in the evening for 14 days (BD+MNT treatment group)
  Interventions: Drug: budesonide
- only intranasal budesonide (Active Comparator): treatment with only intranasal budesonide 1 spray per nostril twice daily for 14 days (BD treatment group)
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — SAR patients received treatment of a combination of budesonide and montelukast tablet or only intranasal budesonide randomly for 14 days
  Other Names: montelukast

SUMMARY:
It is not proven unequivocally whether a combination of an intranasal corticosteroids (INS) and a cysteinyl leukotriene receptor antagonist has greater efficacy than INS in the treatment of severe allergic rhinitis (AR) . We performed a randomized, open-label study in 46 seasonal AR subjects receiving budesonide (BD, 256ug) plus montelukast (MNT, 10 mg) or BD alone (256ug) for 2 weeks. Visual analog scale (VAS) scores, nasal cavity volume (NCV), nasal airway resistance (NAR) and fractional exhaled nitric oxide (FeNO) were assessed before and at end of treatments as the primary treatment outcomes. Similarly, histamine, eosinophil cationic protein (ECP) and cysteinyl-leukotrienes (Cyslts) in nasal secretion and Th1/Th2 cells in nasal mucosa were evaluated as the secondary treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe seasonal allergic rhinitis
* confirmed to had a diagnosis of SAR and also shown to be sensitized to mugwort allergen
* had not received any therapies for AR or antibiotics for at least 7 days before their outpatient clinic visit prior to the study

Exclusion Criteria:

* smokers
* asthma (based on patient's history and pulmonary function tests)
* had any other chronic disease
* pregnant women

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
The change of subjective AR symptoms | at baseline, 14 days
  The participants were asked by one investigator to fill in a questioner detailing the presence of nasal and eye symptoms (including nasal congestion, rhinorrhea, nasal itching, sneezing and eye itching), and to score each symptom on a 0-10 cm scale; with 0 cm = no symptoms and 10 cm = most severe and bothersome symptom. The same investigator calculated both the individual symptom and the average of the sum of 5 AR symptoms scores, before and at the end of 14 days' treatment. Any subject with a mean score of < 4 cm at baseline was excluded from this study.

SECONDARY OUTCOMES:
The change of objective examination: nasal patency | at baseline, 14 days
  Eccovision acoustic rhinometry was used to measure the nasal cavity volume (NCV) according to standardized recommendations. Measurements of nasal volume were made from the first 2 cm (V2), the first 4 cm (V4), from the first 6 cm (V6), from the segment between 0 and 5 cm (V0-5), and the segment between 0 and 7 cm (V0-7) of the nose. All measurements were performed three times by the same operator, and nasal volumes were calculated as the sum of both nostrils24. In the current study, the change in the nasal cavity volume was measured at 2-5 cm, as this seems to be an important variable for mucosal changes.24 Nasal airway resistance (NAR) was measured by anterior active rhinomanometry in a quiet room at temperature of 25°C and humidity of 70%. NAR was measured at 75 Pa point (R75T).
The change of Fractional Exhaled NO | at baseline, 14 days
  A nitric oxide analyser was used to measure exhaled nasal nitric oxide (nNO). Briefly, NO-free air was aspirated through the nasal cavity at a flow rate of 50 ml/s. The subject exhaled against the air-resistance, resulting in an intraoral pressure to close the velum and prevent mixture of oral and nasal gas. Nasal gas from this circuit was continuously routed in part directly into the analyser for determination of nNO, and the level of nNO(ppb) was calculated from a plateau lasting for at least 3s.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Luo, Principal Investigator — Beijing Institute of Otolaryngology
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Price DB, Swern A, Tozzi CA, Philip G, Polos P. Effect of montelukast on lung function in asthma patients with allergic rhinitis: analysis from the COMPACT trial. Allergy. 2006 Jun;61(6):737-42. doi: 10.1111/j.1398-9995.2006.01007.x. PMID 16677244
- [Background] Brozek JL, Bousquet J, Baena-Cagnani CE, Bonini S, Canonica GW, Casale TB, van Wijk RG, Ohta K, Zuberbier T, Schunemann HJ; Global Allergy and Asthma European Network; Grading of Recommendations Assessment, Development and Evaluation Working Group. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines: 2010 revision. J Allergy Clin Immunol. 2010 Sep;126(3):466-76. doi: 10.1016/j.jaci.2010.06.047. PMID 20816182
- [Background] Priftis KN, Drigopoulos K, Sakalidou A, Triga M, Kallis V, Nicolaidou P. Subjective and objective nasal obstruction assessment in children with chronic rhinitis. Int J Pediatr Otorhinolaryngol. 2006 Mar;70(3):501-5. doi: 10.1016/j.ijporl.2005.07.027. Epub 2005 Sep 9. PMID 16154642
- [Background] Henriksen AH, Sue-Chu M, Holmen TL, Langhammer A, Bjermer L. Exhaled and nasal NO levels in allergic rhinitis: relation to sensitization, pollen season and bronchial hyperresponsiveness. Eur Respir J. 1999 Feb;13(2):301-6. doi: 10.1034/j.1399-3003.1999.13b14.x. PMID 10065672
- [Background] Taylor DR, Pijnenburg MW, Smith AD, De Jongste JC. Exhaled nitric oxide measurements: clinical application and interpretation. Thorax. 2006 Sep;61(9):817-27. doi: 10.1136/thx.2005.056093. PMID 16936238
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Clement PA, Gordts F; Standardisation Committee on Objective Assessment of the Nasal Airway, IRS, and ERS. Consensus report on acoustic rhinometry and rhinomanometry. Rhinology. 2005 Sep;43(3):169-79. PMID 16218509